CLINICAL TRIAL: NCT01815658
Title: "Bio-logical" Carbon Fiber Intramedullary Nail Biomechanical Test and Preliminary Clinical Results
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-15-2013
Record Dates: First submitted 2013-03-11; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Broken humerus shaft: Patients presenting with broken humerus shaft
  Interventions: Device: Carbon fiber intramedullary nail (PEEK-CF)

INTERVENTIONS:
Device: Carbon fiber intramedullary nail (PEEK-CF) — Carbon fiber polyether-ether-ketone (PEEK-CF) PICCOLE Nail - produced by Carbofix, Herzlyia, Israel.

SUMMARY:
The aim of this study is to present a novel Intramedullary Nail (IMN) made of CFR - PEED composite, that is biomechanically tailored to closely match cortical bone. This IMN should promote fracture healing and prevent stress shielding osteopenia.

Case records of patients with humurus shaft fracture will be retrospectively reviewed to determine whether the implant promotes bone healing.

ELIGIBILITY:
Inclusion Criteria:

* Broken humerus shaft

Exclusion Criteria:

* All others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with broken humerus
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Bone healing | 6 months
  Observed imaging proof of callus will indicate quality of bone healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel